CLINICAL TRIAL: NCT03836768
Title: A Phase Ib Study of BTK Inhibitor DTRMWXHS-12 in Patients With Relapsed/Refractory Mantle Cell Lymphoma (MCL)
Brief Title: BTK Inhibitor DTRMWXHS-12 in Mantle Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang DTRM Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DTRM_DTRMWXHS-12_004
Record Dates: First submitted 2019-01-30; First posted 2019-02-11 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — DTRMWXHS-12

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Treatment (Experimental): DTRMWXHS-12, oral capsule, daily, 28 days as a cycle
  Interventions: Drug: DTRMWXHS-12

INTERVENTIONS:
Drug: DTRMWXHS-12 — DTRMWXHS-12 capsules: 150 mg, 300 mg

SUMMARY:
The Primary Objective is to evaluate the safety and tolerability of the DTRMWXHS-12 capsule in patients with relapsed/refractory MCL and recommend the dose and dosing method (RP2D) used in phase II study.

The Secondary Objective is to evaluate the pharmacokinetics (PK) of multiple dose oral administration of DTRMWXHS-12 capsule in patients with relapsed/refractory MCL.

The Exploratory Objective is to preliminarily evaluate the efficacy of DTRMWXHS-12 capsule in patients with relapsed/refractory MCL.

ELIGIBILITY:
Inclusion Criteria

1. 18-75 Years old (include 18 and 75), gender is not limited.
2. Measurable lesions by computed tomography (CT)/magnetic resonance imaging (MRI). A measurable lesion is defined as follows: at least the longest diameter of one lymph node >1.5cm and clearly measurable in two vertical directions, or at least the longest diameter of one extranodal lesion >1cm (e.g., liver nodule); If only spleen or gastrointestinal mucosa is involved, corresponding examinations and evaluations will be conducted in the investigator's opinion.
3. The diagnosis report must contain morphology and evidence of positive cyclin D1 by immunohistochemistry or evidence of t (11; 14). The above results are tested by immunohistochemistry, cytogenetics or Fluorescent in situ hybridization (FISH). After enrollment, tumor tissue (FFPE) blocks or sections must be sent to the central laboratory for confirmation of MCL.
4. The laboratory parameters are as follows:

   1. Hematology: Neutrophils ≥ 1.0×10^9/L without growth factor or blood transfusion, platelets ≥ 75×10^9L (≥50×10^9/L if bone marrow is involved), and hemoglobins > 9g/dL within 7 days before enrollment into the study.
   2. Liver: Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) ≤ 2.5×ULN; total bilirubin ≤ 2×ULN (< 3×ULN when diagnosed as Gilbert's syndrome).
   3. Kidney: Creatinine clearance≥30 ml/min (Evaluated by estimated glomerular filtration rate [eGFR] according to the Cockcroft-Gault Equation or the calculation equation of each site); Cockcroft-Gault equation= Female: (140-age)×weight(kg)×0.85/(72×serum creatinine (mg/dL)) Male: (140-age)×body weight(kg)/(72×serum creatinine(mg/dL))
   4. international normalized ratio(INR) ≤ 1.5×ULN and activated partial thromboplastin time (APTT) ≤ 1.5×ULN, and for patients with acquired hemophilia or those treated with clotting factor inhibitors or vitamin K antagonists, the enrollment will be determined after discussion with the investigator.
5. ECOG performance status score 0-2.
6. Life expectancy > 3 months.
7. There must be documentations on relapsed or refractory lymphoma or disease progression after systemic therapy and at least one but less than five therapies for mantle cell lymphoma were administrated previously (1 ≤ number of previous therapies < 5).
8. No response with the last therapy (SD or PD during the treatment), or PD after the therapy.
9. Patients with disease recurrence at least 3 months after autologous hematopoietic stem cell transplantation can be enrolled into the study, if there isn't any relevant active infection.
10. Females of child-bearing potential must agree to use highly effective contraception methods during the study and at least 180 days after the last dose of the investigational drug. Highly effective contraception methods include abstinence, hysterectomy, bilateral ovariectomy without menstruation for six consecutive months, intrauterine contraception systems, hormonal contraception such as injectable contraceptives and oral contraceptives. Males must be sterilized via either vasectomy, or use barrier methods, while their female partners should take the effective contraception methods mentioned above.
11. Patients are voluntary to sign the informed consent form and can understand and comply with all study requirements.

Exclusion Criteria

1. Patients suffering from or previously suffering from CNS lymphoma.
2. Patients received other BTK inhibitors prior to enrollment. Patients who received steroid anti-tumor therapy (a dose equivalent to>20mg/day of prednisone) within 7 days, or received chemotherapy, targeted therapy, or radiotherapy within 4 weeks, or received anti-tumor Chinese medicinal herbs or antibody therapy within 4 weeks, prior to first administration of DTRMWXHS-12 capsule.
3. Patients received major surgery in the past 4 weeks before screening (determined by the investigator according to the patient's condition).
4. Patients with active bleeding or combination with anticoagulant therapy within 3-6 months.
5. Patients had undergone chemotherapy before and in whom the toxicity has not resolved (the toxicity has not resolved to ≤ grade 1 as per National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, except for hair loss, absolute neutrophil count (ANC) and platelets). For neutrophils and platelets, please refer to the criterion 4 [Neutrophils] and [Platelets] in the inclusion criteria.
6. Patients with a history of other active malignant diseases within 2 years prior to enrollment into the study, excluding the following: (1) adequately treated cervical carcinoma in situ; (2) local skin basal cell carcinoma or squamous cell carcinoma; (3) malignant diseases that has been controlled and completely locally treated (by surgery or other means)
7. Patients suffering from active cardiovascular diseases with clinical significance, such as uncontrolled arrhythmia, congestive heart failure, Grade 3 or 4 heart disease according to New York Heart Association (NYHA) Functional Classification, or those with history of myocardial infarction within 6 months before screening.
8. QTcF>450 msecs or other significant ECG abnormalities, including second-degree atrioventricular block type Ⅱ, third-degree atrioventricular block.
9. Patients who can't swallow capsules or with diseases significantly affect the gastrointestinal function, such as malabsorption syndrome, gastric or intestinal resection, symptomatic inflammatory bowel disease, or partial or complete intestinal obstruction.
10. Uncontrolled systemic infections or infections requiring to be treated with intravenous antibacterial agents.
11. Patients who previously received allogeneic stem cell transplantation.
12. Patients known to have been infected with human immunodeficiency virus (HIV) or active hepatitis B or hepatitis C virus (polymerase chain reaction [PCR] or reverse transcription- polymerase chain reaction (RT-PCR) shows positive results).
13. Hepatitis B test includes HBsAg, HBcAb and HBsAb. If the patient is HBsAg-negative but HBcAb-positive (regardless of HBsAb), the PCR technology will be used to detect hepatitis B virus (HBV) DNA, and the acceptable upper limit of normal in the table below is 1000 IU/mL. Considering different PCR kits may be used by different sites, the acceptable upper limit of normal for HBV DNA should be the normal value in the site. Hepatitis C test includes hepatitis C virus (HCV) antibody test, and if the HCV antibody is positive, the RT-PCR technology will be used to detect HCV RNA.
14. Pregnant or lactating women.
15. Any life-threatening disease, medical condition, or organ system dysfunction that, in the investigator's opinion, may affect subject safety or lead to study risks.
16. Patients with poor compliance.
17. Patients who receive treatment with a potent CYP3A (cytochrome P450, family 3, subfamily A) inhibitor or a potent CYP3A inducer within 7 days prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence and severity of (serious) adverse events n each patient according to the NCI-CTCAE4.03 grading | Starting from date of first dose up to 35 days after last dose
  To monitor AEs and SAEs in each patient according to the NCI-CTCAE4.03 grading criteria by evaluating changes in physical examination, laboratory tests, and 12-lead ECG during the whole study

SECONDARY OUTCOMES:
concentration of drug in plasma | From date of first dose to day 56
  concentration of drug in plasma

OTHER OUTCOMES:
Overall response rate (ORR) | From date of first dose to date of disease progression, an average of 6 months
  Percentage of patients with PR, CR

CONTACTS AND LOCATIONS:
Overall Officials: Wei He, Ph.D., Study Director — Zhejiang DTRM Biopharma
Locations (1):
- Peking University Cancer Hospital, Beijing, China